CLINICAL TRIAL: NCT02122432
Title: Impact of Teledermatology Versus Usual Care on Delay Before Diagnosis and/or Treatment of Dermatologic Conditions in General Practice
Brief Title: Teledermatology Versus Usual Care on Delay Before Diagnosis and Treatment of Dermatologic Conditions
Acronym: TELEDERMATO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Paris 7 - Denis Diderot (Other)
Responsible Party: Principal Investigator, TRAN Viet thi, MD, University Paris 7 - Denis Diderot
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DMG002
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Dermatologic Conditions
Keywords: teledermatology; dermatology; general practice; organization of care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teledermatology (Experimental): General practitioner takes 3 photographs per dermatologic lesion using either a telephone with a 3Mega Pixel minimum camera or a standard camera following recommendations of the practice guidelines for teledermatology (2007) of the American Telemedicine Association and sends them to the dermatologist using a secured email server.
  Dermatologist answer is standardized.
  Interventions: Other: Teledermatology
- Usual care (No Intervention): Usual care for dermatologic conditions requiring an expertise from a dermatologist involves the general practitioner 1) giving the patient a paper letter containing at least the following information: date of symptoms, symptomatology, topography of lesions, description of lesions, extension, recent drug intakes) and 2) telling him to see the dermatologist of his choice (patient manages his appointments alone).

INTERVENTIONS:
Other: Teledermatology — General practitioner takes 3 photographs per dermatologic lesion using either a telephone with a 3Mega Pixel minimum camera or a standard camera following recommendations of the practice guidelines for teledermatology (2007) of the American Telemedicine Association.
  Photographs are sent by email using a secured mail server with at least the following information=date of symptoms, symptomatology, topography of lesions, description of lesions, extension, recent drug intakes)
  Photographs are read and analyzed by a single dermatologist who gives an expert answer (diagnosis and/or treatment). Answer is sent back to the general practitioner by email (using a secured mail server). Answer contains at least the following information= are photographs usable? What is the diagnosis? If necessary, which treatment should the general practitioner begin ? If necessary, does the patient need a consultation with a dermatologist ?
  Arms: Teledermatology

SUMMARY:
In France, there is usually a long delay (approximately 6 weeks) before a general practitioner can obtain a specialized advice by dermatologists for diagnosis of "unusual" dermatologic conditions of their patients.

Previous studies have shown that teledermatology is a reliable way for diagnosis in dermatology.

We hypothesize that a teledermatology advice could reduce delay before diagnosis and therefore treatment for patients.

DETAILED DESCRIPTION:
In France, there is usually a long delay (approximately 6 weeks) before a general practitioner can obtain a specialized advice by dermatologists for diagnosis of "unusual" dermatologic conditions of their patients.

Previous studies have shown that teledermatology is a reliable way for diagnosis in dermatology.

We hypothesize that a teledermatology advice could reduce delay before diagnosis and therefore treatment for patients.

ELIGIBILITY:
Inclusion Criteria:

* Consultation with a general practitioner for any motive during which, the general practitioner deems necessary to obtain a dermatologic expertise for a skin lesion (for diagnosis or treatment)

Exclusion Criteria:

* Emergency, assessed by the general practitioner (needs care or quick telephonic advice in the next 24 hours)
* Patients for which diagnosis and/or treatment are known by the general practitioner (the GP needs a dermatologic advice for a specific treatment (for example= laser, instrumental treatment...))
* Patient cannot go the dermatologic consultation by himself (for example: dependant patients...)
* Cognitive or psychiatric impairment (cannot give informed consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Delay before expertise by a dermatologist | 3 months
  Delay, in days, between a patient's consultation with his general practitioner and expertise by a dermatologist (teledermatology or classic consultation) that allows either diagnostic and/or initiation of treatment.
  For example: in the teledermatology group, if the specialist needs to see the patient because the photographs cannot be analyzed correctly, date of expertise is the date of the consultation with the dermatologist.
  Data is censured after 3 months.

SECONDARY OUTCOMES:
Patient's satisfaction | 1 month after expertise by dermatologist
  An investigator will call patients by telephone and assess their satisfaction with their care for the dermatologic condition using a simple rating scale with 4 items ranging from "Not satisfied" (1) to "very satisfied" (4).

OTHER OUTCOMES:
Physicians satisfaction with teledermatology | 3 months
  questionnaire at the end of the study using simple rating scales ranging from "Not satisfied" (1) to "very satisfied" (4)
Number of non usable photographs in teledermatology group | 3 months
  Number of non usable photographs in teledermatology group. Assessment by dermatologists who received the photograph. Reasons for non usability

CONTACTS AND LOCATIONS:
Overall Officials: Viet Thi Tran, MD, Principal Investigator — University paris Diderot
Locations (1):
- University paris Diderot, Paris, France

REFERENCES:
- [Derived] Piette E, Nougairede M, Vuong V, Crickx B, Tran VT. Impact of a store-and-forward teledermatology intervention versus usual care on delay before beginning treatment: A pragmatic cluster-randomized trial in ambulatory care. J Telemed Telecare. 2017 Sep;23(8):725-732. doi: 10.1177/1357633X16663328. Epub 2016 Aug 5. PMID 27496852